CLINICAL TRIAL: NCT00812526
Title: Regulation of Choroidal Blood Flow During Combined Changes in Intraocular Pressure and Arterial Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhöfer, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-190702
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Autoregulation
Keywords: Choroid; Regional blood flow; Autoregulation; Laser Doppler flowmetry

INTERVENTIONS:
Procedure: Suction cup application
Procedure: Squatting

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. For a long time it had been assumed that the choroid is a strictly passive vascular bed, which shows no autoregulation. However, recently several groups have identified some autoregulatory capacity of the choroid. Choroidal autoregulation was first shown in a rabbit model where intraocular pressure (IOP) and arterial blood pressure could be varied independently. In these experiments regulation of choroidal blood flow was not only dependent on ocular perfusion pressure, but was also dependent on the value of IOP. This indicates that a myogenic mechanism contributes to choroidal autoregulation, because the regulatory capacity is dependent on the transmural pressure. In the model of myogenic autoregulation arterioles change their vascular tone depending on the pressure inside the vessel and outside the vessel. The present experiments are designed to test whether a myogenic mechanism may also be involved in choroidal autoregulation in humans. For this purpose the investigators perform experiments during which the IOP and the arterial blood pressure is increased. According to the myogenic theory of autoregulation one would expect stronger vasoconstriction at lower IOPs for the same increase in ocular perfusion pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 1 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Presence of intraocular pathology: ocular hypertension, glaucoma, retinal vasculopathy or other retinal diseases

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2002-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Relationship between ocular perfusion pressure and choroidal blood flow | 4 study days

SECONDARY OUTCOMES:
Choroidal blood flow | 4 study days
Mean arterial pressure | 4 study days
Intraocular pressure | 4 study days
Systolic/diastolic blood pressure | 4 study days

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Polska, MD, Study Director — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria